CLINICAL TRIAL: NCT01928589
Title: Randomized Phase II Study of Partial Breast Irradiation and Sequential vs. Concurrent Chemotherapy in Women With Early Stage Breast Cancer (PBI 3.0)
Brief Title: Partial Irradiation and Sequential vs. Concurrent Chemo Early Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Zellars (Other)
Responsible Party: Sponsor-Investigator, Richard Zellars, Professor and Chairman of the Department of Radiation Oncology, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J13104
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Adenocarcinoma of the Breast
Keywords: Cyclophosphamide; Doxorubicin; Docetaxel; Carboplatin; Herceptin; Partial Breast Irradiation; Concurrent Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Randomized trial of Partial Breast Irradiation (PBI) with concurrent or sequential chemotherapy
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- PBI (Active Comparator): 270 cGy (centigray) x 15
  Interventions: Other: PBI with sequential chemotherapy
- PBI with chemotherapy (Experimental): 270 cGy (centigray) x 15 concurrent with chemotherapy of the treating medical oncologist's choice
  Interventions: Other: PBI with concurrent chemotherapy

INTERVENTIONS:
Other: PBI with sequential chemotherapy — 270 cGy x15
  Other Names: partial breast irradiation with sequential chemotherapy
  Arms: PBI
Other: PBI with concurrent chemotherapy — 270 cGy x15 concurrent with chemotherapy of the treating medical oncologist's choice
  Other Names: partial breast irradiation with chemotherapy
  Arms: PBI with chemotherapy

SUMMARY:
In a small study at Johns Hopkins, women were treated with partial breast irradiation and chemotherapy given at the same time.

We are now testing in a bigger study whether giving partial breast irradiation and chemotherapy at the same time (our new method) has the same side effects and outcomes as giving partial breast irradiation and chemotherapy at different times(older method). In this study women who had their breast cancer removed but need radiation to the breast will be randomized to partial breast irradiation at the same time as chemotherapy or partial breast radiation at a different time than chemotherapy. Randomization is like flipping a coin but in this study about 2 of every 3 women will get the new method.

DETAILED DESCRIPTION:
Breast conserving therapy (BCT) defined as lumpectomy and adjuvant whole breast irradiation (WBI) is integral to the treatment of early stage breast cancer (ESBC). In these patients, BCT provides equivalent survival to mastectomy. Despite equivalent survival, many patients still choose mastectomy over the BCT in light of the 5-7 week commitment required for radiation therapy (XRT). Partial breast irradiation, however, has provided women with ESBC an alternative option for XRT. Worth noting, is PBI offers several advantages over WBI including; decreased duration of XRT, and reduced radiation dose delivery to normal breast tissue and surrounding organs.

Several large trials have advanced the adoption of PBI as a treatment option for women with ESBC. Results of these trials unfortunately differ in regards to patient outcomes. Some trials report no significant difference in the local failure rate (LFR) between intraoperative radiation therapy, interstitial brachytherapy and standard WBI following lumpectomy (Vaidya et al. Lancet 2010; Polgar et al. IJROBP 2004). While others, have demonstrated similar outcomes for PBI and WBI only apply to a select group of patients. (Khan et al. International Journal of Radiation Oncology *Biology *Physics (IJROBP) 2012; Shaitelman et al. Cancer 2010; Stull et al. ASTRO 2012).

A growing body of evidence now suggests, that there is in fact a subgroup of patients for which PBI may not be appropriate. In particular, patients with estrogen receptor (ER) negative tumors have been observed to have higher LFR than patients with ER positive tumors. Stull et al. reported a 3-year LFR of 2% and 12% in ER positive (n=149) and ER negative (n=17) tumors, respectively (Stull et al. ASO 2012). Additionally, Shaitelman et al. reviewed patients treated on the Mammosite registry and found the hazard ratio for local failure was 4.01 in women with ER negative compared to ER positive disease (n=991). (Shaitelman et al. Cancer 2010)

To address the variation in patient outcomes for women treated with PBI, American Society for Radiation Oncology (ASTRO) published a consensus statement grouping patients into "suitable," "cautionary," or "unsuitable" categories. These groupings sought to identify populations best suited for PBI. Patients with ER negative breast cancer were assigned to either the cautionary or unsuitable categories. Shah et al. published a pooled analysis (n=1978) that found the only significant factor associated with ipsilateral breast recurrence (IBRT ) in women who received PBI was ER status. (Shah et al. IJROBP 2012). Leonardi et al. reported similar findings; local recurrence was 2.68 (p = 0.0003) more likely in ER negative (n=189) than in ER positive (n=1608) breast cancers (Leonardi et al. IJROBP 2012). These results suggest that perhaps, patients with ER negative disease are not the most appropriate patients to be treated with PBI.

In addition to radiation therapy, patients are often treated with chemotherapy. Chemotherapy has traditionally been administered either before or after PBI. There are potentially significant benefits, however, that can be gained by the simultaneous administration of chemotherapy and PBI. Administrations of radiation with concurrent chemotherapy soon after surgery will not only shorten the overall duration of therapy, but has the potential to capitalize on the synergy between the two treatment modalities and improve local control. Reports of prohibitive toxicity with concurrent administration of anthracycline-based chemotherapy with WBI have made this approach unpopular. The smaller fields employed during PBI may provide an alternative option. PBI has the potential to reduce toxicity and accelerate the radiation treatment schedule.

To date, we have been able to conduct two phase I trials of PBI and concurrent chemotherapy (PBICC). In both trials we tested whether the toxicity remained prohibitive with this combined treatment regimen. In the first trial, 25 patients were treated with PBI and concurrent dose dense doxorubicin and cyclophosphamide. In the second trial, 34 patients were treated similarly but selection of the chemotherapy regimen was at the discretion of the treating medical oncologist. Results from both trials revealed that PBICC well appears to be tolerated. Specifically, there was no grade 3 or 4 acute or late radiation induced toxicity in either trial. Although these trials were not powered for local failure, one significant finding from these trials was there were no local failures in the first trial (median follow up 6 years), and only one failure (low grade DCIS) in the second trial (median follow up 2.5 years). Interestingly, there were no recurrences in the 21 patients with ER negative tumors or the 17 patients with triple negative tumors.

Our center is the only center to have investigated and published phase I trials of PBICC. Through these trials we have demonstrated preliminary information that PBICC is safe, feasible, and effective treatment option for women with ESBC. Based on our unique experience, we hypothesize that women with ER negative ESBC treated with PBICC will have local control rates similar to women with ER positive disease. Additionally, we hypothesize that women placed in the prone position will have an even more favorable toxicity profile than women placed in the supine position for both PBI and WBI. To further substantiate the low toxicity associated with PBICC and to test this our improved local control hypothesis, we will conduct a randomized prospective trial of PBI with concurrent vs. sequential chemotherapy in women with ER negative or positive ESBC. Our primary endpoint is acute grade 3-4 radiation toxicity and our secondary endpoints will be local control and breast specific quality of life

ELIGIBILITY:
Inclusion Criteria Age ≥ 18 years. Patient must have histologically confirmed (by routine H&E staining) invasive adenocarcinoma of the breast. Primary tumor ≤ 4cm and 0-3 positive axillary lymph nodes (T1-2, N0-1, M0). Margin negative surgery. For subjects with two breasts, they must have had a bilateral mammogram prior to surgery. Patient must have a Medical Oncology consult with the recommendation of chemotherapy. Recommended regimens are as follows: Cyclophosphamide and Doxorubicin (AC); Taxotere, Doxorubicin and Cyclophosphamide (TAC); Taxotere and Cyclophosphamide (TC); or Taxotere, Carboplatin withTrastuzamab (TCH) prior to registration; or Paclitaxel and Trastuzumab. The use of additional chemotherapy, hormonal therapy or Trastuzumab after the initial regimen is at the discretion of the Medical Oncologist. Other primary regimens are possible but the PI must be notified prior to enrollment.

Partial breast irradiation must be scheduled to begin less than 71 days from the last breast surgical procedure. ECOG performance status ≤ 1. Women of child-bearing potential must have a negative (urine or blood) pregnancy test within 6 weeks prior to start of protocol therapy. Women of childbearing potential must also use effective non-hormonal contraception while undergoing radiation treatment and chemotherapy. Note: Women over the age of 70 will not be considered as having child-bearing potential for this study.

Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria Patients who have received neoadjuvant chemotherapy or neoadjuvant hormonal therapy for the current cancer. Patients with squamous cell cancer or sarcomas of the breast. Patients who have active local-regional disease prior to registration. Patient with a prior ipsilateral breast cancer (invasive or non-invasive) from which the patient has been disease free for less than 5 years.

Patient is pregnant. Patient has a serious medical or psychiatric illness which prevents informed consent or adherence with treatment. Study team (PI, Co-I, and or research nurse) may deny enrollment if in the study team's opinion, the candidate may not be adherent to the treatment protocol including scheduled follow-ups.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-01-16 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or 4 short-term toxicity | 6-7 month follow-up
  The primary endpoint will be short term (from baseline to the 6-7 month follow-up) grade 3 or 4 toxicity: confluent moist desquamation, pitting edema, ulceration, hemorrhage or necrosis. Our primary objective is to determine if chemotherapy and PBI can be given concurrently with short term toxicity comparable to standard of care, whole breast radiation (WBR) without chemotherapy, and not inferior to that of PBI plus chemotherapy given sequentially.

SECONDARY OUTCOMES:
1st tumor recurrence | 6-7 months
  Evaluate and compare any first tumor recurrence (local plus distant) between arms of the study.
Long-term grade 3-4 toxicities | Q6-12M 12-18, 24-30, 36-42, 48-54, 60
  Evaluate long term skin toxicity with concurrent chemotherapy and compare between arms of the study.
Time to tumor recurrence | Q6-12M 12-18, 24-30, 36-42, 48-54, 60
  Evaluate and compare Ipsilateral Breast Tumor Recurrence (IBTR), local recurrence, distant recurrence, and disease free survival.
Quantify risks and benefits comparison for each arm | Q6-12M 12-18, 24-30, 36-42, 48-54, 60
  Give a description of the risks and benefits observed in each arm of the study over the duration of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Zellars, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Comprehensive Cancer Center
Locations (10):
- United States (10):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - IU Health Arnett, Lafayette, Indiana
  - John Hopkins University, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Reading Hospital, West Reading, Pennsylvania
  - York Cancer Center, York, Pennsylvania
  - University of Texas-San Antonio, San Antonio, Texas